CLINICAL TRIAL: NCT05508685
Title: Effects of Hiit Associated With Emotional Regulation on Negative Emotions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Irinaldo Capitulino de Souza, principal investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICdesouza
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: High Intensity Exercise; Cognitive Reassessment Strategy
Keywords: High-Intensity Interval Training; Emotional Regulation; Affect
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT and Cognitive Reassessment (Experimental): The experimental group will receive high-intensity interval training associated with cognitive reassessment
  Interventions: Other: HIIT and Cognitive Reassessment
- HIIT Group (Active Comparator): The HITT group will receive only the exercise without cognitive reassessment
  Interventions: Other: HIIT group
- Emotional regulation strategy group (Active Comparator): This group will receive only cognitive reassessment strategy
  Interventions: Other: Emotional regulation strategy group
- Group No exercise and cognitive reassessment (Placebo Comparator): This group will only be evaluated in pre and post, without intervention.
  Interventions: Other: placebo group

INTERVENTIONS:
Other: HIIT and Cognitive Reassessment — Participants will receive 40 minutes of high-intensity interval training focusing on the upper and lower limbs associated with a cognitive reassessment strategy during the exercises.
  Arms: HIIT and Cognitive Reassessment
Other: HIIT group — Participants will receive high-intensity interval training, lasting 40 minutes, focusing on upper and lower limbs.
  Arms: HIIT Group
Other: Emotional regulation strategy group — Participants will be instructed to cognitively reassess the negative emotions they feel or do not feel during the practice of the exercises. Participants will receive instructions on how to reassess.
  Arms: Emotional regulation strategy group
Other: placebo group — Participants in this group will not receive any intervention. Only pre and post experiment will be evaluated.
  Arms: Group No exercise and cognitive reassessment

SUMMARY:
Despite the benefits of physical exercise, the population does not adhere to the recommended levels of physical activity. The reported difficulties in starting and maintaining a physical exercise program are attributed to personal barriers and lack of motivation. Thus, there is an urgent need for efficient intervention proposals to increase engagement in daily physical exercise. High-intensity interval training (HIIT) is a promising and economical method, aiming at the development of efforts at high, maximum or supramaximal intensity, based on several methods: calisthenics (using the body's own strength) resistance (heavy objects, bars or devices for high-repetition resistance activities) and traditional (exercise modalities such as running and cycling). Emotional regulation (ER) is essential for the psychosocial well-being of human beings and is defined as the ability to influence, experience and express emotions, being an action, conscious or not, that directly modulates emotions and alters their nature as the intensity and duration. Regular physical exercise has been attributed to a reduction in depression symptoms, an increase in emotional well-being and a reduction in negative feelings. In addition to physical exercise, the use of cognitive reassessment to regulate emotions was positively associated with a decrease in negative affect in psychopathological diagnoses.

DETAILED DESCRIPTION:
Main goal

To evaluate the effects of high-intensity interval training (HIIT) associated with a cognitive reassessment strategy on negative emotions in sedentary women.

Specific objectives

Evaluate and compare the positive and negative affective of women in three moments; Evaluate and compare the intensity and valence of emotions in three moments; Investigate possible associations between emotion dysregulation and emotion regulation strategies in positive and negative affect; Investigate and compare HIIT intensity and emotion regulation strategy in pleasure and displeasure during physical exercise during practice.

ELIGIBILITY:
Inclusion criteria:

• No psychiatric or neurological disorder

Exclusion criteria:

* Using mood-altering medications
* Joint problems
* Practicing physical activity for six months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Affect Scale | Fifteen days
  Each item is rated on a five-point Likert scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely, to measure the extent to which affect was experienced in a specified period of time.

SECONDARY OUTCOMES:
Self Assessment Manikin | Fifteen days
  The Self-Assessment Mannequin (SAM) is a non-verbal pictorial assessment technique that directly measures pleasure, arousal, and mastery associated with a person's affective reaction to a wide variety of stimuli. The reports are subjective to measure a series of images that varied in both valence and affective intensity.
Feeling Scale | Fifteen days
  The feeling scale was used to assess affective valence. The 11-point bipolar scale ranging from very bad (-5) to very good (+5), with anchors at Neutral (0) and all odd integers, including bad (-3), fairly bad (-1), reasonably good (+1) and good (+3).
The Perceived Effort Scale | Fifteen days
  Borg's Perceived Exertion Rating (RPE) is a way of measuring the intensity level of physical activity. These include a rating of 6 perceiving "no exertion" to 20 perceiving a "maximum exertion" of exertion. Practitioners generally agree that perceived exertion ratings between 12 and 14 on the Borg Scale suggest that physical activity is being performed at a moderate level of intensity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dryman MT, Heimberg RG. Emotion regulation in social anxiety and depression: a systematic review of expressive suppression and cognitive reappraisal. Clin Psychol Rev. 2018 Nov;65:17-42. doi: 10.1016/j.cpr.2018.07.004. Epub 2018 Jul 23. PMID 30064053
- [Background] Edwards MK, Rhodes RE, Mann JR, Loprinzi PD. Effects of acute aerobic exercise or meditation on emotional regulation. Physiol Behav. 2018 Mar 15;186:16-24. doi: 10.1016/j.physbeh.2017.12.037. Epub 2018 Jan 5. PMID 29309746
- [Background] Evans, M., Rohan, K. J., Howard, A., Ho, S. Y., Dubbert, P. M., & Stetson, B. A. (2017). Exercise dimensions and psychological well-being: A community-based exercise study. Journal of Clinical Sport Psychology, 11(2), 107-125.